CLINICAL TRIAL: NCT03364218
Title: Nebulized N-Acetyl Cysteine for Bronchiolitis in Inpatient Hospital Use: A Randomized Controlled Trial
Brief Title: Nebulized N-Acetyl Cysteine for Bronchiolitis in Inpatient Hospital Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Rahul Pandey, Assistant Professor, Pediatric Critical Care Medicine, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB# 2314
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Bronchiolitis Acute
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Subjects will receive N-Acetyl Cysteine (NAC) nebulized 2 mL of 10% NAC solution every 12 hours during their stay in the Pediatric Intensive Care Unit.
  Interventions: Drug: N-Acetyl Cysteine
- Control Group (No Intervention): Subjects will not receive NAC, but will receive standard care for acute bronchiolitis.

INTERVENTIONS:
Drug: N-Acetyl Cysteine — Nebulized N-Acetyl Cysteine administered every 12 hours
  Other Names: NAC
  Arms: Treatment Group

SUMMARY:
Bronchiolitis is the major cause of hospital admission in infants < 6 months of age and usually viruses like Respiratory syncytial virus (RSV), human metapneumo virus, Adeno virus, para-influenza virus, Rhino virus and influenza virus are the main culprit. In the US, acute bronchiolitis in infancy is responsible for approximately 150,000 hospitalizations yearly at an estimated cost of $500 million. Globally in 2005 it was estimated that at least 33.8 million were affected with RSV and in the same year, RSV associated severe acute lower respiratory infection (ALRI) were responsible for ~3.4 million hospitalizations and 66,000-199,000 deaths worldwide, with 99% of these deaths in developing countries.

In acute bronchiolitis there is cellular swelling and excessive mucus production. There is also proliferation of goblet cells, which leads to increased mucus production. The excess mucus produced is poorly cleared by non-ciliated (regenerating) epithelial cells leading to areas of narrowing and blocking of the bronchioles, causing the airway obstruction, hyperinflation, increased airway resistance, atelectasis and increased ventilation-perfusion mismatch that characterize acute bronchiolitis.

Currently there is no medicine that has proven effective in treating acute bronchiolitis and per American Academy of Pediatrics guidelines the management of acute bronchiolitis remains supportive care for the acute respiratory failure associated with acute bronchiolitis.

N-Acetyl Cysteine (NAC) is an antioxidant, anti-mucus compound that increases intracellular glutathione at the cellular level. It cleaves disulfide bonds by converting them to two sulfhydryl groups. This action results in the breakup of mucoproteins in lung mucus, reducing their chain lengths and thinning the mucus. Nebulized NAC is not studied well in acute bronchiolitis and is uncommonly used for the same. NAC has been studied in the treatment of various disease states, including those pulmonary in nature such as cystic fibrosis, chronic bronchitis, non-cystic fibrosis bronchiectasis and found to be beneficial.

With this background knowledge, the purpose of this study is to evaluate the effectiveness of nebulized mucolytic therapy in treatment of children with viral bronchiolitis.

DETAILED DESCRIPTION:
A randomized clinical trial with blinding of person assigned for assessing and scoring the patients. The participants will include children less than 2 yrs. age admitted to the Pediatric Intensive Care Unit (PICU) with a diagnosis of acute bronchiolitis who will be randomized into either the NAC group or the non-NAC (Control) group.

Patients with acute bronchiolitis who require to be started on high flow nasal cannula support or any other noninvasive ventilator/BIPAP support are transferred/directly admitted to PICU. There is no time limit between when patients are admitted and when patients must sign consent or be randomized.

After a patient with acute bronchiolitis is identified, a member of the study team will perform a chart review to assess eligibility as described by the inclusion/exclusion criteria. If eligible, parent(s)/guardian(s) will be approached and Informed Consent will be obtained. Using randomization software(www.randomizer.org) the enrolled patients will be randomly assigned to either the NAC group or the non-NAC (Control) group.

The NAC will be ordered by the on call pharmacist and it will be administered by the on call Respiratory therapists. Between the two groups only the NAC group will get nebulized 2 ml of 10% NAC solution every 12 hours during their stay in PICU.

The PICU uses HHFNC (humidified high flow nasal canula), Heliox and non-invasive ventilation such as RAM canula, Neurally adjusted ventilatory assist (NAVA) and BIPAP. The PICU also typically uses Dexmedetomidine infusion once the patient is on non invasive ventilation (NIV) as a light sedation medication to avoid agitation and better ventilation patient synchrony.

The scoring tool used by Seattle children's Bronchiolitis pathway will be used. HHFNC (humidified high flow nasal cannula) will be started for patients when scores are ≥2. Depending on the clinical worsening the patient may require help with Heliox and escalation to non-invasive ventilation.

There will be twice a day blind assessments completed by experienced PICU/Transport nurses who were non-involved in patient care in PICU at that time. The pharmacist is going to use randomization software to randomly assign patients to a group (i.e control vs treatment). Also, the pharmacist will order code called as "Trial***" in the medical record (*** denotes a number assigned) and depending on the randomization the patient may or may not get the trial medication (Nebulized NAC). As such, all patients in the study will have a medical record orders which look similar to help achieve blinding at this stage for the treating physicians and independent evaluators.

All patients in the study will receive a type of respiratory support, such as High flow nasal cannula, noninvasive ventilator/ BIPAP etc. and because the NAC neb can easily be given through those circuits, no extra equipment will be required for patients who are in the treatment (NAC) group. Given that there is no difference in equipment in both treatment and control groups, the only way the double-blind is broken in this scenario is NAC's odor.

The odor of Neb NAC typically stays in the room during the treatment (2-3 minutes) and should not last >30 minutes after every administration. NAC is a sulfur compound and hence smells like "rotten eggs" so for precaution to maintain blindness, a respiratory therapist will spray a commercial rotten egg smelling solution at approximately the same time as treatment is administered for all patients in the study.

Because the NAC neb will be delivered through a closed respiratory circuit and also because the respiratory therapists use filters for nebulization treatments, the chances of sticky residues will be lower and hence difficult to figure out by examination.

The 12 hourly neb treatments will occur from 6:30-7:30am and pm respectively. This timing works in favor for blinding because both attending physicians and the independent evaluators are less likely to be present during this time. The assessment will involve scoring the patients according to the bronchiolitis scoring data tool. These assessments will be completed for the duration of the PICU stay. The on service PICU attendings will only be involved in clinical management of patients and will be blinded from randomization. The blinding will be broken if one of the on service physicians or PICU/Transport nurses performing assessments are aware of the currently admitted patient randomization details.

Reasons subjects may be withdrawn from the study: patient gets transferred to another facility due to family's requests, family wishes to withdraw in the middle of the study, or to protect the welfare of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Full term new born neonates up to patients < 2yrs
* Respiratory score ≥2
* Otherwise healthy with new respiratory illness

Exclusion Criteria:

* Prematurity <34 weeks for patients <6 months age.
* h/o congenital heart disease requiring baseline medication
* Patient received diagnosis of Asthma or reactive airway disease in past.
* Anatomic airway defect.
* Immunodeficiency
* Chronic lung disease
* Patients who have had previous bronchiolitis < 4 weeks ago
* Patients intubated for acute bronchiolitis during the current admission.
* h/o Larynogomlacia, bronchomalacia or tracheomalacia.

Ages: 1 Week to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Score | 1. Twice daily by physician 2. 15-30 min pre-treatment by nurse 3. 15-30 and 90 min post-treatment by nurse
  4 item scoring system completed by clinician used to assess respiratory symptoms. Each item is scored 0-3, with the value increasing as severity of symptoms increases.
Time on Non-Invasive Ventilation | From time of PICU admission to time of PICU discharge, assessed up to 4 weeks
  Length of time on NIV
Duration of PICU/Hospital Admission | From time of hospital admission to time of hospital discharge, assessed up to 4 weeks
  Length of time patient remains hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Pandey, MD, Principal Investigator — Carilion Medical Center
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No